CLINICAL TRIAL: NCT03900234
Title: Cross-Sectional Population Based Study on Prevalence and Risk Factors for Chronic Venous Disease in General Population
Brief Title: Prevalence of Chronic Venous Disease in General Population
Status: Completed | Type: Observational
Sponsor: Pirogov Russian National Research Medical University (Other)
Responsible Party: Principal Investigator, Igor Zolotukhin, Professor, Pirogov Russian National Research Medical University
Other Study IDs: 15
Record Dates: First submitted 2019-03-29; First posted 2019-04-02 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-04

CONDITIONS: Chronic Venous Insufficiency
Keywords: chronic venous disease; prevalence; risk factors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Residents of the single rural settlement: No interventions will be administered
  Interventions: Other: No intervention will be administered

INTERVENTIONS:
Other: No intervention will be administered — No intervention will be studied. Clinical and ultrasound examinations will be used to find the prevalence of CVD.

SUMMARY:
This study is designed to find prevalence and risk factors for chronic venous disease (CVD) in the general population. All the resident, who live in a single rural settlement will be invited to participate.

DETAILED DESCRIPTION:
The study has cross-sectional design. All the residents aged 10 and more, living in the single rural settlement located in Central Russia will be invited to participate in the study.

Those who agree, will be examined both clinically and by duplex ultrasound. Medical history of participants will be taken, demographic data will be collected. Possible factors that may influence CVD development will be registered.

Signs and symptoms of CVD will be registered. Duplex ultrasound will be used in every resident to reveal pathological venous reflux in deep and superficial veins.

ELIGIBILITY:
Inclusion Criteria:

* residents living in the rural settlement where study will be conducted
* both female and male
* age 10 years and more
* agree to participate
* signed infromed consent

Exclusion Criteria:

* age 9 years and less
* not signed informed consent

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All the residents of 10 years and more living in the same settlement, willing to participate will be included
Sampling Method: Non-Probability Sample
Enrollment: 783 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2015-08-31 (Actual); Study Completion 2015-08-31 (Actual)

PRIMARY OUTCOMES:
Presence of chronic venous disease | up to Sept. 2015
  As a disease positive subjects with any morphological and functional abnormalities of the venous system of long duration manifested either by symptoms and/or signs indicating the need for investigation and/or care will be considered

CONTACTS AND LOCATIONS:
Overall Officials: Igor Zolotukhin, Prof, Principal Investigator — Russian National Research Medical University
Locations (1):
- Pirogov Russian National Research Medical University, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No
No IPD are going to be shared with other researchers

REFERENCES:
- [Derived] Zolotukhin IA, Seliverstov EI, Shevtsov YN, Avakiants IP, Tatarintsev AM, Kirienko AI. Risk factors for venous symptoms in Russian patients with chronic venous disease. Curr Med Res Opin. 2019 Sep;35(9):1583-1587. doi: 10.1080/03007995.2019.1605050. Epub 2019 May 13. PMID 30958033